CLINICAL TRIAL: NCT00821236
Title: A Prospective, Multi Center Clinical Comparison of Fellow Eyes Undergoing Lasik Using the Wavelight Allegretto Wave™ Excimer Laser in One Eye and the Amo/Visx Customvue™ or the Ladarvision 4000 Excimer Laser System in the Contralateral Eye
Brief Title: Contralateral Comparison of Three Excimer Laser Systems in Performing LASIK
Acronym: WLCVLV-001
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Durrie Vision (Other)
Collaborators: Alcon Research (Industry)
Responsible Party: Principal Investigator, Daniel S. Durrie, MD, President, Durrie Vision
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WLCVLV-001
Record Dates: First submitted 2009-01-09; First posted 2009-01-13 (Estimated); Results first posted 2013-03-01 (Estimated); Last update posted 2013-03-01 (Estimated); Status verified 2013-01

CONDITIONS: Myopia; Astigmatism
Keywords: Myopia; LASIK; Astigmatism; Laser Vision Correction; Excimer Laser
MeSH Terms: conditions — Myopia; Astigmatism | interventions — Lasers, Excimer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Wavelight (Active Comparator): WaveLight ALLEGRETTO WAVE™ wavefront guided or optimized excimer laser treatment
  Interventions: Device: Excimer Laser
- AMO/VISX CustomVue (Active Comparator): AMO/VISX CustomVue™
  Interventions: Device: AMO/VISX CustomVue™
- LADARVision 4000 excimer laser (Active Comparator): LADARVision 4000 excimer laser
  Interventions: Device: LADARVision 4000 excimer laser

INTERVENTIONS:
Device: Excimer Laser — WaveLight ALLEGRETTO WAVE™ wavefront guided or optimized excimer laser treatment
  Arms: Wavelight
Device: AMO/VISX CustomVue™ — Excimer Laser
  Arms: AMO/VISX CustomVue
Device: LADARVision 4000 excimer laser — Excimer Laser
  Arms: LADARVision 4000 excimer laser

SUMMARY:
The purpose of this study is to compare LASIK outcomes using the WaveLight ALLEGRETTO WAVE™ wavefront guided or optimized excimer laser treatment with the AMO/VISX CustomVue™ and the LADARVision 4000 excimer laser treatment.

Standard refractive outcomes such as uncorrected and best corrected visual acuity, and intended vs. achieved postoperative refractions will be evaluated; in addition, high order optical aberrations, contrast sensitivity, and topography will be measured.

DETAILED DESCRIPTION:
The primary objective of this study is to compare WaveLight ALLEGRETTO WAVE™ wavefront guided or optimized excimer laser treatment with the AMO/VISX CustomVue™ and the LADARVision 4000 excimer laser treatment using both subjective and objective outcome measures. This comparison will be made between fellow eyes of the same patient following excimer laser ablation using the WaveLight ALLEGRETTO WAVE™ Excimer Laser System in one eye and the AMO/VISX CustomVue™ or the LADARVision 4000 excimer laser in the contralateral eye .

ELIGIBILITY:
Inclusion Criteria:

* Subjects who have up to -7.00D of spherical equivalent myopia or myopia with astigmatism, with up to -7.00D of spherical component and up to 3.00 D of astigmatic component at the spectacle plane in both eyes.
* Subjects must have a stable refraction as documented by previous clinical records. Spherical equivalent has not progressed at a rate of more than 0.50D per year prior to the baseline examination in both eyes or as documented by clinical judgment by the investigator.
* Subjects who wear contact lenses must discontinue wear at least 3 days for soft and at least 3 weeks for RGP prior to the preoperative evaluation or surgery, in either eye.
* Subjects must have visual acuity correctable to at least 20/20 in both eyes.
* Subjects must be at least 18 years of age.
* Subjects must be willing and able to return for scheduled follow up examinations for twelve months after LASIK surgery.
* Subjects must sign and be given a copy of the written Informed Consent form.

Exclusion Criteria:

* Subjects for whom both eyes do not meet all inclusion criteria and either eye meets any exclusion criteria.
* Subjects for whom the combination of their baseline corneal thickness and the planned operative parameters for the LASIK procedure would result in less than 250 microns of remaining posterior corneal thickness below the flap postoperatively in either eye.
* Eyes for which the baseline standard manifest refraction exhibits greater than 1.00D more minus in sphere power, or a difference of greater than 0.75 D in cylinder power.
* Subjects desiring spherical under correction in one eye (i.e. no monovision correction is permitted).
* Subjects for whom the preoperative assessment of the ocular topography and /or aberrations indicates that either eye is not a suitable candidate for LASIK vision correction procedure. Examples include frank or forme frust keratoconus, corneal warpage, pellucid marginal degeneration, etc.
* Subjects with clinically significant dry eye syndrome or clinically significant blepharitis in either eye.
* Subjects with anterior segment pathology, including clinically significant cataracts or corneal scarring or neovascularization in either eye.
* Subjects with residual, recurrent, active ocular or eyelid disease, including any corneal abnormality (specifically, recurrent corneal erosion, severe basement membrane disease) in either eye.
* Subjects with ophthalmoscopic signs of progressive or unstable myopia or keratoconus (or keratoconus suspect) in either eye.
* Subjects with unstable (distorted/not clear) corneal mires on central keratometry in either eye.
* Subjects who have undergone previous intraocular or corneal surgery of any kind, including any type of surgery for either refractive or therapeutic purposes in either eye.
* Subjects who have a history of Herpes zoster or Herpes simplex keratitis.
* Subjects on chronic systemic corticosteroid or other immunosuppressive therapy that may affect wound healing, any immunocompromised subjects, and subjects with clinically significant atopic disease, connective tissue disease, or diabetes.
* Subjects with a history of steroid-responsive rise in intraocular pressure, glaucoma, or preoperative Intraocular pressure>23 mm Hg in either eye.
* Subjects with macular pathology in either eye.
* Subjects who are pregnant, lactating, or planning to be pregnant during the course of the study.
* Subjects with known sensitivity to planned study concomitant medications.
* Subjects participating in any other ophthalmic drug or device clinical trial during the time of this clinical investigation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2009-01; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel S. Durrie, MD, Principal Investigator
Locations (2):
- United States (2):
  - Durrie Vision, Overland Park, Kansas
  - Karl G. Stonecipher, MD, Greensboro, North Carolina

RESULTS

PARTICIPANT FLOW:
Groups:
- Lasik for Treatment of Nearsightedness: WaveLight ALLEGRETTO WAVE™ wavefront guided or optimized excimer laser treatment LADARVision 4000 excimer laser AMO/VISX CustomVue™ excimer laser treatment
Period: Overall Study
Arm/Group | Lasik for Treatment of Nearsightedness
Started | 40
Completed | 37
Not Completed | 3
Not completed — Lost to Follow-up | 3

BASELINE CHARACTERISTICS:
Groups:
- LADARVision 4000 Excimer Laser: LADARVision 4000 excimer laser treatment
- Total: Total of all reporting groups
Arm/Group | Wavelight | AMO/VISX CustomVue | LADARVision 4000 Excimer Laser | Total
Number analyzed (Participants) | 20 | 10 | 10 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 20 | 10 | 10 | 40
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 6 | 6 | 25
  Male | 7 | 4 | 4 | 15

OUTCOME MEASURES:

1. Primary Outcome: 1 Day Postoperative Lasik Uncorrected Visual Acuity
Description: Visual acuity measured without glasses or contact lenses. LogMar is a method of measuring visual acuity. Generally speaking, the U.S. population is familiar with 20/20 visual acuity reference. Samples of LogMar equivalent values would be 20/20=0.0 LogMar, 20/25=0.1 LogMar, 20/16=-0.1, etc.
Time Frame: 1 Day
Measure: Mean (Standard Deviation); unit: LogMar
Arm/Group | Wavelight | AMO/VISX CustomVue | LADARVision 4000 Excimer Laser
Number analyzed (Participants) | 20 | 10 | 10
LogMar | -0.04 (0.08) | -0.05 (0.06) | 0.06 (0.16)

2. Primary Outcome: 1 Week Postoperative Lasik Uncorrected Visual Acuity
Description: Visual acuity measured withouth glasses or contact lenses. LogMar is a method of measuring visual acuity. Generally speaking, the U.S. population is familiar with 20/20 visual acuity reference. Samples of LogMar equivalent values would be 20/20=0.0 LogMar, 20/25=0.1 LogMar, 20/16=-0.1, etc.
Time Frame: 1 week post op
Measure: Mean (Standard Deviation); unit: LogMar
Arm/Group | Wavelight | AMO/VISX CustomVue | LADARVision 4000 Excimer Laser
Number analyzed (Participants) | 20 | 10 | 10
LogMar | -0.04 (5.27) | -0.09 (2.36) | -0.02 (5.8)

3. Primary Outcome: 1 Month Postoperative Lasik Visual Acuity
Description: as for outcome 1
Time Frame: 1 Month Postoperative
Measure: Mean (Standard Deviation); unit: LogMar
Arm/Group | Wavelight | AMO/VISX CustomVue | LADARVision 4000 Excimer Laser
Number analyzed (Participants) | 20 | 10 | 10
LogMar | -0.1 (0.09) | -0.11 (0.06) | 0.08 (-0.08)

ADVERSE EVENTS:
Arm/Group | Wavelight | AMO/VISX CustomVue | LADARVision 4000 Excimer Laser
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/20 | 0/10 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No